CLINICAL TRIAL: NCT01357967
Title: The Effect of Quetiapine XR in Depressive Patients Showing Aberrant N100 Amplitude Slope
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Inje University (Other)
Responsible Party: Principal Investigator, Seung-Hwan Lee, Professor, Inje University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Seroquel ISS D1443C00053
Record Dates: First submitted 2011-05-19; First posted 2011-05-23 (Estimated); Last update posted 2012-11-01 (Estimated); Status verified 2012-10

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Quetiapine Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Seroquel XR adjunctive (Experimental): The quetiapine XR adjunct group will be titrated up to 300mg. Initial dosing will begin at 50mg on Day 1 and 2, increased to 150mg on Day 3 and 4. Further adjustments will be able to be made upwards or downwards within the recommended dose range of 50mg to 300mg depending upon the clinical response and tolerance of the patient. Seroquel XR will be administered daily in the evening.
  The dosage of SSRIs will be maintained as low (es-citalopram 5mg, paxil CR 6.25mg, fluoxetine 10mg, and sertraline 25mg).
  Interventions: Drug: Seroquel XR adjunctive
- SSRI monotherapy (Active Comparator): active comparator
  Interventions: Drug: SSRI monotherapy

INTERVENTIONS:
Drug: SSRI monotherapy — SSRI (paxil CR, es-citalopram, fluoxetine, sertraline) start with (paxil CR 12.5mg, es-citalopram 10mg, fluoxetine 20mg, sertraline 50mg) for 1 week up to maximal dosage, flexible dosage, usually in the morning
  Other Names: SSRI
  Arms: SSRI monotherapy
Drug: Seroquel XR adjunctive — Quetiapine group:
  seroquel XR 50mg Day 1 --> 50mg Day 2 --> 150mg Day 3 --> 150mg Day 4 --> adjustment usually at hs but can be daytime
  Other Names: Seroquel XR; quetiapine XR; quetiapine
  Arms: Seroquel XR adjunctive

SUMMARY:
Recently, there are increasing data about intensity dependent amplitude change (IDAP: N100 amplitude slope) of auditory evoked Event Related Potential (ERP) components for its role on surrogate marker of central serotonergic activity. A high N100 amplitude slope reflects low serotonergic neurotransmission and vice versa. There are a couple of studies reporting associations of N1 amplitude slope with response to Citalopram (positive correlation) and Reboxetine (negative correlation) treatment in major depressive disorder patients (2,3). The investigator also published a case series about SSRI super-sensitivity and SSRI induced mania in patients with aberrantly high N100 slope (4). And serotonin transporter gene polymorphism was studied for its role about pathophysiology of bipolar disorder (5, 6, 7). Serotonin promoter gene was known to have significant relationship with N100 amplitude slope (8). Furthermore previous study showed that N100 amplitude slope was well correlated with hypomanic and hyperthymic personality (9).

Conclusively from above results, the investigator hypothesized that if depressive patients show aberrant high or low N100 amplitude slope (N100 response outliers), they will not response well to SSRI medication. They will response better to quetiapine XR adjunctive therapy. In this study, the investigator will confirm it by comparing treatment effect between SSRI monotherapy and quetiapine XR adjunctive in aberrant N100 responder.

Hypothesis First visit depressive patients might have monopolar or bipolar depression. If depressive patients show aberrantly high or low N100 amplitude slope, they will not response to SSRI medication.

Patients who have aberrantly high or low N100 amplitude slope will response better to quetiapine XR adjunctive therapy.

DETAILED DESCRIPTION:
1.2 Rationale for this study The development of better strategy for treatment of major depressive disorder and other mood disorder is a very important issue for patients, mental health provider and government. So far, treatments of depressive illness have been based on mainly trial and error method and physician's personal experiences.

So the development of new strategy for predicting better treatment response group of quetiapine XR would be great contributions for basic brain science and mental health fields.

2. STUDY OBJECTIVES

2.1 Primary objective

Primary target of this study is to prove the following hypothesis :

Patients who have aberrantly high or low N100 amplitude slope will response better to quetiapine XR adjunctive therapy.

2.2 Secondary objectives

Patients who have aberrantly high or low N100 amplitude slope will show higher dropout rate for SSRI monotherapy compared to quetiapine XR adjunctive.

3. STUDY PLAN AND PROCEDURES

3.1 Overall study design and study plan

This study will be conducted by open, randomized, two armed, and observational phase IV study. The investigator will compare treatment response between Quetiapine XR and SSRIs to major depressive disorder patients showing aberrant response of N100 amplitude slope. The investigator will use SSRIs drugs (paxil CR, es-citalopram, fluoxetine, sertraline) as comparator drug. The investigator will recruit drug naive patients but if there were previous antidepressant medication, washout periods will be required for one week. This study will be conducted as single centre study, and patients will be enrolled based on the DSM-IV major depressive disorder criteria, and also aberrant response of N100 amplitude (N100 slope < 0.21, or > 1.59, this criteria can be revised base on our newly published data). In and out-patients status of patients will recruited together. The treatment duration will be six weeks from beginning of pharmacological treatment.

Procedure for measuring the LDAEP (N100 amplitude slope)

Recording took place in an electrically shielded and sound attenuated room adjacent to the recording apparatus (Synamps, Neuroscan ®). Subjects were seated with open eyes in a slightly reclined chair with a head rest. Evoked responses were recorded with 32 electrodes referred to Cz. Pure sinus tones (1000 Hz, 80 ms duration with 10 ms rise and 10 ms fall time, ISI randomized between 500 and 900 ms) of 5 intensities (55, 65, 75, 85, 95 dB sound pressure level) were presented binaurally in a pseudo-randomised form by audiometry headphones. Data were collected with a sampling rate of 1000 Hz and an analogous bandpass filter (1-30 Hz). Analysis was performed with the Scan® software package version 4.3. One hundred ms prestimulus and 300 ms poststimulus periods were evaluated for about 100 sweeps of every intensity (all together 500 sweeps). For artifact suppression, all trials were automatically excluded from averaging, if the voltage exceeded ± 70uV in any one of the 32 channels at any time point of the averaging period. For each subject, the remaining sweeps were averaged separately for the five stimulus intensities. At least 30 artefact-free sweeps/intensity had to be averaged. N1 peaks (80-140 ms) and P2 peaks (100-250 ms) were determined semi-automatically at the Cz electrode (referred to linked-mastoids). The IDAP was calculated as linear regression slope with stimulus intensity as independent and N1/P2 amplitude as dependent variable.

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the study patients must fulfill all of the following criteria:

1. Major depressive disorder (HRDS > 18)
2. N100 amplitude slope outlier (< 0.21 or > 1.59)
3. Aged 18 to 55 years
4. Provision of written informed consent prior to any study specific procedures

Exclusion Criteria:

Any of the following is regarded as a criterion for exclusion from the study:

1. Pregnancy or lactation: : urine HCG (-)
2. Any DSM-IV Axis I disorder not defined in the inclusion criteria
3. Patients who, in the opinion of the investigator, pose an imminent risk of suicide or a danger to self or others
4. Known intolerance or lack of response to quetiapine fumarate and SSRI antidepressant, as judged by the investigator
5. Hearing impairment
6. Use of any of the following cytochrome P450 3A4 inhibitors in the 14 days preceding enrollment including but not limited to: ketoconazole, itraconazole, fluconazole, erythromycin, clarithromycin, troleandomycin, indinavir, nelfinavir, ritonavir, fluvoxamine and saquinavir
7. Use of any of the following cytochrome P450 3A4 inducers in the 14 days preceding enrollment including but not limited to: phenytoin, carbamazepine, barbiturates, rifampin, St. John's Wort, and glucocorticoids
8. Administration of a depot antipsychotic injection within one dosing interval (for the depot) before randomisation/baseline
9. Substance or alcohol dependence at enrollment (except dependence in full remission, and except for caffeine or nicotine dependence), as defined by DSM-IV criteria
10. Opiates, amphetamine, barbiturate, cocaine, cannabis, or hallucinogen abuse by DSM-IV criteria within 4 weeks prior to enrollment
11. Medical conditions that would affect absorption, distribution, metabolism, or excretion of study treatment
12. Unstable or inadequately treated medical illness (e.g. congestive heart failure, angina pectoris, hypertension or clinically relevant abnormal laboratory values) as judged by the investigator
13. Involvement in the planning and conduct of the study
14. Previous enrollment or randomisation of treatment in the present study.
15. Participation in another drug trial within 4 weeks prior enrollment into this study or longer in accordance with local requirements
16. A patient with Diabetes Mellitus (DM) fulfilling one of the following criteria

    * Unstable DM defined as enrollment glycosylated hemoglobin (HbA1c) > 8.5%
    * Admitted to hospital for treatment of DM or DM related illness in past 12 weeks.
    * Not under physician care for DM
    * Physician responsible for patient's DM care has not indicated that patient's DM is controlled.
    * Physician responsible for patient's DM care has not approved patient's participation in the study
    * Has not been on the same dose of oral hypoglycaemic drug(s) and/or diet for the 4 weeks prior to randomisation. For thiazolidinediones (glitazones) this period should not be less than 8 Weeks.
    * Taking insulin whose daily dose on one occasion in the past 4 weeks has been more than 10% above or below their mean dose in the preceding 4 weeks Note: If a diabetic patient meets one of these criteria, the patient is to be excluded even if the treating physician believes that the patient is stable and can participate in the study.
17. An absolute neutrophil count (ANC) of <= 1.5 x 1,000,000,000 per liter

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-05; Primary Completion 2012-12 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in HDRS scale | 0,1,2,4,6 weeks
  -Hamilton Depression Rating Scale (HDRS) : Baseline, 1, 2, 4, 6 week

SECONDARY OUTCOMES:
Change from baseline in CGI, BDI, and YMRS scales | 0,1,2,4,6 weeks
  * Clincal Global Impression (CGI) : Baseline, 1, 2, 4, 6 week
  * Beck Depression Inventory (BDI) : Baseline, 1, 2, 4, 6 week
  * Young Mania rating Scale (YMRS) : Baseline, 1, 2, 4, 6 week

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Hwan Lee, MD, PhD, Principal Investigator — Psychiatry Department Inje University Ilsan Paik Hospital
Locations (2):
- South Korea (2):
  - Psychiatry Department, Inje University Ilsan Paik Hospital, Goyang, Geyonggi
  - Inje University Ilsanpaik Hospital, Goyang-si, Gyeonggi-do